CLINICAL TRIAL: NCT02432196
Title: Safety and Performance Study of the Harpoon Medical Transapical Suturing Device (TSD-5) in Subjects With Degenerative Mitral Regurgitation - CE Mark Study for the Harpoon Medical Device in Poland
Brief Title: CE Mark Study for the Harpoon Medical Device in Poland
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Edwards Lifesciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HMFIM -1000-PL-04
Record Dates: First submitted 2015-04-27; First posted 2015-05-04 (Estimated); Results first posted 2019-11-25 (Actual); Last update posted 2024-01-22 (Actual); Status verified 2024-01

CONDITIONS: Mitral Valve Regurgitation; Mitral Valve Prolapse; Mitral Valve Insufficiency
Keywords: Mitral Valve Repair; Transapical; artificial chordae
MeSH Terms: conditions — Mitral Valve Insufficiency; Mitral Valve Prolapse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Harpoon Medical TSD-5 (Experimental): This is a prospective, nonrandomized, single-centered European study designed single arm study to demonstrate the performance and safety of the Harpoon Medical TSD-5 in Subjects with degenerative mitral regurgitation.
  Interventions: Device: Harpoon Medical Device

INTERVENTIONS:
Device: Harpoon Medical Device — It is expected that the Harpoon Medical transapical suturing device will be a valuable treatment alternative for patients suffering from mitral valve regurgitation because it can access the left ventricle with a small shaft or via a small valved introducer with a secure anchoring mechanism that can be deployed anywhere on the mitral valve leaflet.

SUMMARY:
The purpose of this study is to evaluate the safety and performance of the Harpoon Medical TSD-5. The Harpoon device will provide many significant advantages over current surgical interventions including: 1) a small minimally invasive incision, 2) no sternotomy, 3) no cardiopulmonary bypass, 4) no aortic manipulation, 5) a direct path to the valve plane, 6) performed on a beating heart, 7) real-time TEE-guided chordal length adjustment and 8) less complicated procedure that is teachable and adoptable.

DETAILED DESCRIPTION:
The TSD-5 is intended to secure ePTFE sutures on the mitral valve for the treatment of mitral valve disease.

ELIGIBILITY:
Inclusion Criteria:

* All subjects referred for mitral valve surgery
* Presence of severe mitral regurgitation as read on an echocardiographic study performed within 60 days prior to procedure. Assessment of mitral regurgitation will be performed by the investigational site echocardiography laboratory and confirmed by the Core Echocardiography Laboratory using an integrative method.
* Age > 18 years
* Estimated post-ePTFE cordal implantation coaptation surface is adequate in the judgment of the operating surgeon and the patient eligibility committee
* Degenerative mitral valve disease
* Subject is able to sign informed consent and able to return for follow-up and is capable of participating in all testing associated with this clinical investigation
* Women of child-bearing potential have a negative pregnancy test
* Able to sign informed consent

Exclusion Criteria:

* Age < 18 years
* Infective endocarditis
* Anterior or bileaflet prolapse
* Functional mitral regurgitation
* History of Mediastinal Radiation
* Inflammatory (rheumatic) valve disease
* Requirement for concomitant cardiac surgery (e.g., coronary artery bypass grafting (CABG), aortic valve surgery, etc.)
* Symptomatic coronary artery disease
* Cardiogenic shock at the time of enrollment
* ST segment elevation myocardial infarction requiring intervention within 30 days prior to enrollment
* Evidence of cirrhosis or hepatic synthetic failure
* Pregnancy at the time of enrollment (women of child bearing age should have negative pregnancy within 14 days of surgery)
* Severe pulmonary hypertension (PA systolic pressure > 70 mmHg)
* Previous cardiac surgery, or surgery on the left pleural space
* Left ventricular, atrial or appendage thrombus
* Severely calcified mitral leaflets
* Recent stroke (< 6 months) with permanent impairment
* EuroScore (for mitral valve repair) > 8%
* Subjects with contraindications to transesophageal echocardiography
* Severe left or right ventricular dysfunction
* NYHA Class IV
* Renal insufficiency CKD stage 3b or worse (GFR < 45 ml/min/1.73 m2)
* Patient is participating in another clinical study for which follow-up is currently ongoing. (Co-enrollment in an investigational device or interventional study)
* Patient with non-cardiac co-morbidities and life expectancy < 1 year
* Patient has a condition or conditions that, in the opinion of the Investigator, preclude participation, including willingness to comply with all follow-up procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2015-12-11 (Actual); Primary Completion 2018-02-08 (Actual); Study Completion 2022-11-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boguslaw Kapelak, MD, PhD, Principal Investigator — John Paul II University Hospital; Piotr Kolsut, MD, PhD, Principal Investigator — Instytut of Kardiologii & Transplantology
Locations (2):
- Poland (2):
  - John Paul II University Hospital, Krakow
  - Instytut of Kardiologii & Transplantology, Warsaw

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be available to other researchers.

REFERENCES:
- [Result] Gammie JS, Wilson P, Bartus K, Gackowski A, Hung J, D'Ambra MN, Kolsut P, Bittle GJ, Szymanski P, Sadowski J, Kapelak B, Bilewska A, Kusmierczyk M, Ghoreishi M. Transapical Beating-Heart Mitral Valve Repair With an Expanded Polytetrafluoroethylene Cordal Implantation Device: Initial Clinical Experience. Circulation. 2016 Jul 19;134(3):189-97. doi: 10.1161/CIRCULATIONAHA.116.022010. PMID 27436878
- [Derived] Gammie JS, Bartus K, Gackowski A, Szymanski P, Bilewska A, Kusmierczyk M, Kapelak B, Rzucidlo-Resil J, Duncan A, Yadav R, Livesey S, Diprose P, Gerosa G, D'Onofrio A, Pittarello D, Denti P, La Canna G, De Bonis M, Alfieri O, Hung J, Kolsut P, D'Ambra MN. Safety and performance of a novel transventricular beating heart mitral valve repair system: 1-year outcomes. Eur J Cardiothorac Surg. 2021 Jan 4;59(1):199-206. doi: 10.1093/ejcts/ezaa256. PMID 33038223
- [Derived] Goto Y, Funada A, Goto Y. Duration of Prehospital Cardiopulmonary Resuscitation and Favorable Neurological Outcomes for Pediatric Out-of-Hospital Cardiac Arrests: A Nationwide, Population-Based Cohort Study. Circulation. 2016 Dec 20;134(25):2046-2059. doi: 10.1161/CIRCULATIONAHA.116.023821. Epub 2016 Oct 24. PMID 27777278

RESULTS

PARTICIPANT FLOW:
Groups:
- Harpoon Medical Device: Safety and Performance study of the Harpoon Medical Device in patients with degenerative mitral regurgitation.
Period: Overall Study
Arm/Group | Harpoon Medical Device
Started (Enrolled in Study) | 26
Completed | 20
Not Completed | 6
Not completed — Exit - did not receive study device | 1
Not completed — Death | 2
Not completed — Reoperation | 3

BASELINE CHARACTERISTICS:
Population: Subjects who had an attempt to be treated with the Harpoon Medical Device.
Groups:
- Harpoon Medical Device: Safety and Performance study of the Harpoon Medical Device in subjects with degenerative mitral regurgitation.
Arm/Group | Harpoon Medical Device
Number analyzed (Participants) | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.2 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 21
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Subject's Procedural Success During the First 30 Days
Description: Procedural success was defined as the patient leaving the operating room with a successful implant of one or more ePTFE cords on the mitral valve and reduced mitral regurgitation from severe to </=moderate at the conclusion of the procedure and at 30 days post-procedure.
Time Frame: Procedure through 30 days
Population: This outcome is reported for subjects who were enrolled in the trial.
Measure: Count of Participants; unit: Participants
Arm/Group | Harpoon Medical Device
Number analyzed (Participants) | 26
Participants | 24

2. Primary Outcome: Percentage of Subject's With Freedom From Serious Adverse Events (SAE) </= 30 Days
Description: Subject's freedom from Serious Adverse Events during the ePTFE implantation procedure and at 30 days follow-up. Time to events were estimated by Kaplan-Meier method.
Time Frame: Procedure through 30 days
Population: This outcome is reported for subjects who were enrolled in the trial where data is available.
Measure: Number; unit: percentage of subjects
Arm/Group | Harpoon Medical Device
Number analyzed (Participants) | 26
percentage of subjects
  KM estimate: Implant | 96.2
  KM estimate: 1 Month | 76.9

3. Primary Outcome: Subject's Serious Adverse Events (SAE) Through Discharge
Description: Number of Participants experiencing a Serious Adverse Event (SAE) through time of Discharge.
Time Frame: Discharge, an average of 6 days post implant
Population: This outcome is reported for subjects who were enrolled in the trial where data is available.
Measure: Count of Participants; unit: Participants
Arm/Group | Harpoon Medical Device
Number analyzed (Participants) | 26
Participants | 4

4. Secondary Outcome: Subject's Severity of Mitral Regurgitation Over Time
Description: Valvular regurgitation occurs when the valve in the heart does not close tightly allowing some of the blood that was pumped out of the heart to leak back into it. Valvular regurgitation is evaluated by echocardiography over time. It is assessed on a scale from 0 to 4, where 0 represents no regurgitation and 4 represents severe regurgitation. The numbers on the scale are reflected as follows: 0 = no leak, 1 = a trace leak, 2 = a mild leak, 3 = a moderate leak, and 4 = a severe leak.
  Higher numbers on the scale show a worsening outcome.
Time Frame: 6 months, 12 months, 18 months, 24 months, 30 months, and 36 months
Population: This outcome is reported for subjects who were enrolled in the trial where data is available.
Measure: Count of Participants; unit: Participants
Arm/Group | Harpoon Medical Device
Number analyzed (Participants) | 26
Participants
  6 month follow-up: number analyzed (Participants) | 23
  6 month follow-up: None | 0
  6 month follow-up: Trace | 13
  6 month follow-up: Mild | 7
  6 month follow-up: Moderate | 2
  6 month follow-up: Severe | 1
  12 month follow-up: number analyzed (Participants) | 21
  12 month follow-up: None | 1
  12 month follow-up: Trace | 13
  12 month follow-up: Mild | 4
  12 month follow-up: Moderate | 3
  12 month follow-up: Severe | 0
  18 month follow-up: number analyzed (Participants) | 4
  18 month follow-up: None | 0
  18 month follow-up: Trace | 3
  18 month follow-up: Mild | 1
  18 month follow-up: Moderate | 0
  18 month follow-up: Severe | 0
  24 month follow-up: number analyzed (Participants) | 19
  24 month follow-up: None | 1
  24 month follow-up: Trace | 13
  24 month follow-up: Mild | 2
  24 month follow-up: Moderate | 3
  24 month follow-up: Severe | 0
  30 month follow-up: number analyzed (Participants) | 8
  30 month follow-up: None | 0
  30 month follow-up: Trace | 6
  30 month follow-up: Mild | 0
  30 month follow-up: Moderate | 2
  30 month follow-up: Severe | 0
  36 month follow-up: number analyzed (Participants) | 13
  36 month follow-up: None | 0
  36 month follow-up: Trace | 8
  36 month follow-up: Mild | 3
  36 month follow-up: Moderate | 2
  36 month follow-up: Severe | 0

5. Secondary Outcome: Percentage of Subject's With Freedom From Serious Adverse Events (SAE) Post-implant > 30 Days
Description: Subject's freedom from Serious Adverse Events at >30 days post-implant. Time to events were estimated by Kaplan-Meier method.
Time Frame: 6 months, 12 months, 18 months, 24 months, 30 months, and 36 months
Population: This outcome is reported for subjects who were enrolled in the trial where data is available.
Measure: Number; unit: percentage of subjects
Arm/Group | Harpoon Medical Device
Number analyzed (Participants) | 26
percentage of subjects
  KM estimate: 6 months | 73.1
  KM estimate: 12 months | 65.4
  KM estimate: 18 months | 53.8
  KM estimate: 24 months | 46.2
  KM estimate: 30 months | 34.6
  KM estimate: 36 months | 34.6

ADVERSE EVENTS:
Time Frame: Events occurring from baseline through 60 months post implant.
Description: Adverse event table is reported for patients who were enrolled in the trial.
Arm/Group | Harpoon Medical Device
All-Cause Mortality (participants affected / at risk) | 2/26
Serious Adverse Events (participants affected / at risk) | 17/26
Other Adverse Events (participants affected / at risk) | 20/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Harpoon Medical Device (N=26)
Arrhythmia - Persistent atrial fibrillation (Cardiac disorders) | 4 (4)
ePTFE cordal rupture (Product Issues) | 4 (4)
Nonspecific, unknown, or other body system - Other complication (General disorders) | 1 (1)
Biliary (gallbladder) (Gastrointestinal disorders) | 1 (2)
Aortic dissection (Cardiac disorders) | 1 (1)
CARDIOVASCULAR - OTHER (Cardiac disorders) | 1 (1)
Bleeding - Gastrointestinal lower - Major (Blood and lymphatic system disorders) | 1 (1)
Bone fracture/Break (General disorders) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1)
Development of regurgitation as a result of technical errors (Product Issues) | 2 (2)
Endocarditis (Cardiac disorders) | 1 (1)
Muscular skeletal/Dermatologic - Other (General disorders) | 2 (2)
Pericardial tamponade (Cardiac disorders) | 1 (1)
Pleural effusion - Left (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sternal wound/Thoracic infection (General disorders) | 1 (1)
MYOCARDIAL INFARCTION (Cardiac disorders) | 1 (1)
RENAL FAILURE - CHRONIC (Renal and urinary disorders) | 1 (1)
VASCULAR - DEEP VEIN THROMBOSIS (DVT) (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Harpoon Medical Device (N=26)
Nonspecific, unknown, or other body system - Other complication (General disorders) | 10 (10)
Arrhythmia - Paroxysmal Atrial Fibrillation (PAF) (Cardiac disorders) | 3 (6)
Muscular skeletal/Dermatologic - Other (General disorders) | 3 (3)
Arrhythmia - Bradycardia (Cardiac disorders) | 2 (2)
Anemia - Bleeding related - Minor (Blood and lymphatic system disorders) | 1 (1)
Arrhythmia - Tachy-bradycardia (Cardiac disorders) | 1 (1)
Bleeding - Pulmonary/Respiratory - Minor (e.g. hemothorax) (Blood and lymphatic system disorders) | 1 (1)
Cardiovascular - Other (Cardiac disorders) | 2 (2)
Damage to the native mitral valve apparatus Chord (Product Issues) | 1 (1)
Hypertension - Systemic (Cardiac disorders) | 3 (4)
Renal dysfunction (Renal and urinary disorders) | 1 (1)
BLEEDING - CARDIOVASCULAR - MINOR (Blood and lymphatic system disorders) | 1 (1)
ANGINA, STABLE (Cardiac disorders) | 1 (1)
PERICARDITIS (Cardiac disorders) | 1 (1)
THROMBOEMBOLIC EVENT - STROKE (Cardiac disorders) | 1 (1)
EPTFE CORDAL RUPTURE (Product Issues) | 1 (1)
GASTROINTESTINAL - OTHER (Gastrointestinal disorders) | 2 (2)
GENITOURINARY - OTHER (Renal and urinary disorders) | 1 (1)
URINARY TRACT INFECTION (UTI) (Renal and urinary disorders) | 1 (1)
ALLERGIC REACTION - OTHER (General disorders) | 1 (1)
CANCER - NEWLY DIAGNOSED (General disorders) | 1 (1)
RESPIRATORY INFECTION - UPPER (URI) (Respiratory, thoracic and mediastinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI must submit publication 60 days prior to its submission for presentation/publication to Sponsor. The Sponsor may, at its sole discretion, (a) approve the publication, (b) reject the publication, or (c) suggest changes to the publication to ensure protection of confidential commercial information in compliance with regulatory requirements. Until the content of any publication is approved by the Sponsor and the PI, the PI shall not disclose such publication.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-07): https://cdn.clinicaltrials.gov/large-docs/96/NCT02432196/Prot_SAP_001.pdf